CLINICAL TRIAL: NCT00453661
Title: Cancer Prevention and Treatment Demonstration for Hispanic Medicare Eligible Beneficiaries - CMS
Brief Title: Cancer Prevention and Treatment Demonstration for Ethnic and Racial Minorities
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2006-0419; CMS-5036-N (Other Grant/Funding Number: Centers for Medicare& Medicaid Services); NCI-2014-02518 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Cervical Cancer; Prostate Cancer; Colorectal Cancer; Lung Cancer
Keywords: Breast Cancer; Cervical Cancer; Prostate Cancer; Colorectal Cancer; Lung Cancer; Cancer Prevention; Treatment Demonstration for Ethnic and Racial Minorities; Centers for Medicare and Medicaid Services; CMS; Hispanic American; Cancer Screening Assessment; Annual Questionnaire; Patient Navigator; Educational Materials
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms | interventions — Surveys and Questionnaires; Patient Navigation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Patient Navigator (PN) + Educational Materials + Annual Questionnaires
  Interventions: Behavioral: Questionnaire; Behavioral: Patient Navigator (PN)
- Comparison Group: Educational Materials + Exit Questionnaire
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Intervention Group:
  Cancer Screening Assessment (CSA) questionnaire 45-60 minutes annually for 4 years + Exit Questionnaire at end of study.
  Comparison Group:
  Exit Questionnaire only.
  Other Names: Survey
Behavioral: Patient Navigator (PN) — Staff member, called patient navigator (PN), who assist with medical care and/or screenings, questionnaires.
  Groups: Intervention Group

SUMMARY:
The goal of this behavioral research study is to improve the use of cancer prevention services, increase early detection, and treatment of cancer. A secondary outcome of this demonstration project proposes that a structured patient navigator (PN) will reduce the cost of Medicare services.

DETAILED DESCRIPTION:
Screening Questionnaire:

Before you can start on this study, you will answer a 20 minute Triage questionnaire. The questionnaire will ask you if you have had cancer, what type of cancer, and when you were last treated.

Cancer-Screening Groups and Treatment Groups:

Once you answer the Triage questionnaire and if you are found to be eligible to take part in this study, you will be placed in the Cancer Screening Group or the Treatment Group based on your answers to the Triage questionnaire.

If you have not been treated for cancer in the past or if it has been more than 5 years since you were last treated, you will be in the Cancer Screening Group and you will complete the screening Cancer Screening Assessment (CSA). The CSA will ask you about cancer screenings, lifestyle, and other health related items. The questionnaire should take about a total of 45-60 minutes to complete.

If you have been treated for cancer in the past 5 years, you will be in the Treatment Group. The CSA will ask you about cancer screenings, cancer treatment, and other health related items. The questionnaire should take about a total of 45-60 minutes to complete.

After completion of the Cancer Screening Assessment (CSA) for either the Cancer Screening Group or the Treatment Group, you will complete a CSA addendum questionnaire. This CSA addendum questionnaire will ask you about barriers and factors that may influence your health related decisions. The questionnaire should take 15-20 minutes to complete.

Intervention and Comparison Groups:

Participants in either the cancer-screening group or the treatment group will be randomly assigned (as in the flip of a coin) to one of 2 additional groups, the "Intervention group" or the "Comparison" group. You will have an equal chance of being in either group.

If you are in the Intervention Group, you will work with a staff member, called a patient navigator (PN), who will assist with medical care and/or screenings (intervention group). For example, the staff member may help schedule screening appointments, medical care appointments, or any other necessary assistance to meet health care needs. The PN will be responsible for recording information about your care and any cancer treatment, should that be necessary.

You will complete a CSA questionnaire 1 time a year for up to 4 years. A staff member will contact you by phone to set up an appointment to give you the CSA questionnaires. All questionnaires will be completed at a time and place that you and the study staff agree upon. For example, the study staff may meet you at a community center, independent-living center, or another agreed upon location. The questionnaire should take about 45-60 minutes to complete.

If you are in the Comparison Group, you will not work with a staff member and you will not complete any additional questionnaires during the 4 years on study.

Both the intervention group and the comparison group will receive educational materials.

Exit Questionnaire:

About 4 years after you join the study, you will be contacted by a staff member and you will set up an exit questionnaire meeting. This questionnaire will be completed at a time and place that you and the staff member agree upon. This questionnaire will contain similar questions to those you have been answering since your participation in the study. The questionnaire will take about 45-60 minutes to complete.

Length of Study:

You will be considered off-study after 4 years.

This is an investigational study. Up to 11,964 participants will take part in this study. A total of 2,812 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must have Medicare Part A and Part B
2. All participants must be Latino / Hispanic American
3. All participants must be at least 40 years of age
4. All Cancer Screening Group participants must be a Medicare-eligible beneficiary from Region 6 (Central Gulf Coast) as defined by Texas Department of State Health Services.
5. All Cancer Treatment Group participants must have been diagnosed with breast, cervix, prostate, colorectal, and/or lung cancer within the past 5 years.
6. All Cancer Treatment Group participants must be a Medicare-eligible beneficiary from Texas.

Exclusion Criteria:

1. All participants must not be enrolled in a managed care plan (also called an HMO, Medicare + Choice, or Medicare Advantage)
2. All participants must not be enrolled in hospice
3. All Cancer Screening Group participants must not have been diagnosed with cancer within the last 5 years.
4. All Cancer Treatment Group participants must not be a Medicare-eligible beneficiary outside of Region 6 (Central Gulf Coast) unless treated at MD Anderson.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hispanic American 40 Years + treated for cancer and Medicare eligible.
Sampling Method: Non-Probability Sample
Enrollment: 2472 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Screening Rates | 4 Years

SECONDARY OUTCOMES:
Compliance Rate Across 5 Cancer Types | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Torres, DRPH,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org